CLINICAL TRIAL: NCT04905732
Title: Nasal High-frequency Oscillatory Ventilation (NHFOV) vs Nasal Continuous Positive Airway Pressure(NCPAP) for Ventilated Newborn Infants With BPD: a Randomized Controlled Trial
Brief Title: Nasal High-frequency Oscillatory Ventilation (NHFOV) for Ventilated Newborn Infants With BPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Collaborators: Children's Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Chen Long,MD, director, Children's Hospital of Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NHFOV for sBPD
Record Dates: First submitted 2021-02-26; First posted 2021-05-28 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Bronchopulmonary Dysplasia; Nasal High-frequency Oscillatory Ventilation; Nasal Continuous Positive Airway Pressure; Neonate
MeSH Terms: conditions — Bronchopulmonary Dysplasia

STUDY DESIGN:
Intervention Model Description: After documenting parental consent, the ventilated infants with BPD were randomly assigned to either NHFOV or NCPAP
Who Masked: Investigator, Outcomes Assessor
Masking Description: After documenting parental consent, these ventilated infants with BPD were randomly assigned to either NHFOV or NCPAP using a table of random numbers and sealed opaque envelopes when they were eligible for extubation. Blinding to doctor was not possible due to the nature of the intervention, is not necessary to participant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NHFOV (Experimental): After documenting parental consent, the ventilated infants with BPD were randomly assigned to NHFOV
  Interventions: Device: NHFOV
- NCPAP (Active Comparator): After documenting parental consent, the ventilated infants with BPD were randomly assigned to NCPAP
  Interventions: Device: NCPAP

INTERVENTIONS:
Device: NHFOV — After documenting parental consent, the ventilated infants with BPD were randomly assigned to NHFOV
  Arms: NHFOV
Device: NCPAP — After documenting parental consent, the ventilated infants with BPD were randomly assigned to NCPAP
  Arms: NCPAP

SUMMARY:
Invasive ventilation(IV) remains one key cornerstone to reduce neonatal mortality for preterm infants with respiratory distress syndrome(RDS) and/or acute respiratory distress syndrome(ARDS). However, it is also related to increased risks of ventilator-associated lung injury and escalation of pulmonary inflammation, and which finally result in bronchopulmonary dysplasia (BPD). Early weaning from IV in newborn infants with BPD is therefore a key procedure to reduce these risks above.

DETAILED DESCRIPTION:
Supplying with the combined advantages of NCPAP and high-frequency oscillatory ventilation (HFOV) with high carbon dioxide(CO2) removal, no need for synchronisation, non-invasion, less volume/barotraumas, and increased functional residual capacity, nasal HFOV(NHFOV) was considered as a strengthened version of NCPAP. Furthermore, the superimposed oscillations of NHFOV could avoid gas-trapping, and allowed to obviously up-regulate mean airway pressure (MAP) more than NCPAP. Thus, NHFOV might be more beneficial as post-extubation respiratory support strategy to avoid re-intubation and subsequent complications and/or sequelae as compared with NCPAP in preterm infants. Nowadays, NHFOV was increasingly used in neonatal intensive care unit (NICU) around the world due to its convenient operation. A retrospective review has reported the beneficial effects of NHFOV in preterm infants as a remedial measure after failing to other noninvasive modes, including reducing the number of apneas, bradycardias or oxygen desaturations. However, there were rare randomized controlled studies comparing NHFOV with NCPAP in preterm infants with BPD.

We have found that NHFOV is superior to NCPAP in avoiding re-intubation in very preterm infants with the first extubation. The purpose of the present study was to compare NHFOV with NCPAP as post-extubation respiratory support strategies on the need for endotracheal ventilation, as well as pressure of CO2(PCO2) level in preterm infants with BPD.

ELIGIBILITY:
Inclusion Criteria:

Eligibility requirements for neonates:

* The gestational age is less than 32 weeks
* The preterm neonates are diagnosed with BPD and need invasive ventilation
* Extubation and subsequent noninvasive ventilation is ready to be carried out

Exclusion Criteria:

one of the following conditions is needed:

* there were no intraventricular hemorrhage(IVH) grades 3 or 4
* major congenital anomalies
* parents' decision not to participate

Ages: 28 Days to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2021-05-20 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
re-intubation rate | seven days after extubation
  the newborn infants with ventilated BPD is reintubated after extubation
death | seven days after extubation
  the newborn infants with BPD die
the level of carbon dioxide | seven days after extubation
  the level of carbon dioxide is measure after extubation between groups

SECONDARY OUTCOMES:
necrotizing entercolitis(NEC) | seven days after extubation
  the newborn infants with BPD is diagnosed with NEC
intraventricular hemorrhage(IVH) | seven days after extubation
  the newborn infants with BPD is diagnosed with NEC

CONTACTS AND LOCATIONS:
Locations (1):
- Chen（陈）, Chongqing, Chongqing Municipality, China